CLINICAL TRIAL: NCT04652791
Title: A Study to Assess Efficacy and Safety of Wangbi Capsule in Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Director, Devision of Rheumatology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 20201005V1
Record Dates: First submitted 2020-11-12; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wangbi Capsule: Patients who are taking Wangbi Capsule for the treatment.
- Other drugs: Patients who are not taking Wangbi Capsule for the treatment.

SUMMARY:
The aim of this multi-center, prospective, non-interventional cohort study is to evaluate the efficacy and safety of Wangbi capsule for rheumatoid arthritis patients in the real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of RA as defined by the ACR/EULAR 2010 classification criteria
* Patients older than 18
* Syndrome of insufficiency of liver and kidney or syndrome of cold and dampness defined by traditional Chinese medicine

Exclusion Criteria:

* Patients who are pregnant or breast feeding at enrolment
* History of malignancy prior to screening
* Patients with severe or poorly controlled chronic diseases such as hypertension, diabetes and coronary heart disease
* Patients taking biological agents, > 10mg prednisone (or equivalent amount of other glucocorticoids) ，more than 2 kinds of DMARDs or similar TCM drug like Wangbi Capsule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Disease Activity Score 28（DAS 28）≤3.2 | Week 52
  Percentage of Participants achieving Disease Activity Score 28（DAS 28）≤3.2 at week 52

SECONDARY OUTCOMES:
Percentage of Participants Achieving American College of Rheumatology Response 20/50/70 | Week 12, Week 24,Week 52
  ACR responders are participants with at least 20%, 50% and 70% improvement from baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: Health Assessment Questionnaire-Disability Index (HAQ-DI) which measures participants perceived degree of difficulty performing daily activities, acute phase reactant as measured by hsCRP, Patient's Assessment of Pain-Visual Analog Scale (Pain-VAS), Patient's Global Assessment of Disease Activity (PaGADA_VAS), and Physician's Global Assessment of Disease Activity (PhGADA_VAS).
Change from baseline in Disease Activity Score Based on 28-Joint Count (DAS28) | Baseline, Week 12, Week 24, Week 52
  DAS28 consists of a composite score of the following variables: tender joint count out of 28 (TJC28), swollen joint count out of 28 (SJC28), hsCRP [milligrams per liter (mg/L)], and Patient's Global Assessment of Disease Activity (PaGADA_VAS) on a 0 to 100 millimeter (mm) VAS (0=very well to 100=very poor). A decrease in DAS28-CRP indicates an improvement in participant's condition.
Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) | Baseline, Week 12, Week 24,Week 52
  The disability assessment component of the HAQ assesses a subjects level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities.
Change From Baseline in erythrocyte sedimentation rate(ESR) | Baseline, Week 12, Week 24,Week 52
  Change From Baseline in erythrocyte sedimentation rate at Week 12，24 and 52
Change From Baseline in C-reactive protein(CRP) | Baseline, Week 12, Week 24,Week 52
  Change From Baseline in C-reactive protein at Week 12，24 and 52
Percentage of Participants Achieving Disease Activity Score 28≤3.2 | Week 12, Week 24
  Percentage of Participants achieving Disease Activity Score 28≤3.2 at week 12 and 24

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China